CLINICAL TRIAL: NCT04760002
Title: Danish Patients With Atrial Fibrillation and Sleep Apnea Prevalence by Night Owl
Acronym: DANAPNO
Status: Completed | Type: Observational
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Morten Lamberts, MD, PhD, Associate professor, Consultant Cardiology,, Herlev and Gentofte Hospital
Other Study IDs: P-2021-57
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation Patients: Atrial fibrillation patients are to be investigated for sleep apnea by the a home-monitoring device.
  Other inclusion criteria are:
  >18 years <90 years
  Interventions: Device: NightOwl

INTERVENTIONS:
Device: NightOwl — The NightOwl consists of a small sensor device which is placed on the fingertip and a smartphone app that is connected to an encrypted cloud-based analytics platform within the European Union, the NightOwl software. It is self-applied by attaching the sensor to the fingertip by means of an adhesive patch. The NightOwl sensor acquires accelerometer data and reflectancebased photoplethysmography (PPG) from which it derives actigraphy (sleep/wake behavior), SpO2, peripheral artery tone (PAT) and pulse rate, among other features. A PAT analysis derives changes in caliber of arteries elicited by alterations in the contractile activity of vascular smooth muscle and are referred to as changes in arterial tone. The end state of the apnea-hypopnea events are associated with sympathetic activation.

SUMMARY:
A project of the feasibility of using NightOwl to detect the prevalence of obstructive sleep apnea (OSA) in patients with atrial fibrillation (AF). The long-term aim is to use the device to screen for OSA in a randomized clinical trial in AF patients undergoing ablation and/or a randomized trial of AF patients undergoing cardioversion.

DETAILED DESCRIPTION:
Patients diagnosed with any type of AF referred to anticoagulation initiation at a nurse-run ambulatory will beasked to participate. The ambulatory consists of four daily nurse-led tracks at Department ofCardiology, Herlev-Gentofte University Hospital. In a formal collaboration, Department ofPulmonology, Herlev-Gentofte University Hospital provides work-up with cardio-respiratory monitoring investigation and clinical evaluation of initiating treatment of sleep apnea in patients referred from the study. ParticipantsParticipants with AF, without known sleep apnea, and indication for anticoagulation will be recruited from the Thrombosis unit (Tromboseklinikken) at Herlev-GentofteHospital. Participants will be contacted and asked of participation in the research project by a local investigator or a project nurse as part of their standard check at the anticoagulation outpatient clinic at Herlev and Gentofte Hospital. The conversation will include verbal participant information about the research project and about the right of time to consider recruitment. The written participant information will be handed to the participants prior to the verbal information, and it will be handed to the participants by a researcher with thorough knowledge to the project or a project nurse. The information needed for finding qualified participants, before a written informed consent is obtained, will be passed on to the investigators. The written informed consent allows the researchers to obtain necessary information for the project in the participant's medical health records

Study Design:

The is a cross sectional study. In total two visits will be planned, with a third visit for the first 20 participants and participants with apnea-hypopnea index (AHI)>15 included in the study.

1. Initial visit with time for clinical evaluation, questionnaire of OSA symptoms, theparticipant borrows a NightOwl and receive device instructions.
2. Four night of recording with NightOwl™ in home environment.
3. Follow-up visit for the home-monitoring results and soft node questionnaire.
4. For the 20 first patients and for all patients where the home test is showing (AHI>15) a fourth visit at the sleep apnea clinic will be arranged.

The time plan for the study inclusion until last patient enrolled are estimated to be approximately 6months

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AF of any type
2. Age < 90 years
3. Age >18 years

Exclusion Criteria:

1. Known sleep apnea
2. Secondary AF (post-surgical, due to infection, thyroid-induced)
3. Known or newly discovered severe ventricular ectopic beats (as defined by the NightOwl manual)
4. Professional drivers
5. Severe heart failure (New York Heart Association class III or IV)
6. Severe chronic obstructive pulmonary disease (use of home oxygen)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with AF referred to anticoagulation initiation at a nurse-run ambulatory will be asked to participate.
  Participants will be recruited from the Thrombosis unit (Tromboseklinikken) at Herlev-Gentofte Hospital. Patient reporting of symptoms for sleep apnea is not included as inclusion or exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea in atrial fibrillation patients | 6 months
  The primary outcome of the study is the prevalence with 95% confidence intervals of obstructive sleep apnea in atrial fibrillation patients detected by NightOwl.

SECONDARY OUTCOMES:
Correlation between NightOwl and cardio-respiratory monitoring | 6 months
  The secondary outcome will be correlation between NightOwl and cardio-respiratory diagnostic testing for obstructive sleep apnea and correlation between obstructive sleep apnea screening questionnaire for cardio-respiratory and NightOwl.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev-Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen MH, Dalgaard F, Laub RR, Gottlieb V, Hansen ML, Vendelboe O, Hansen J, Lamberts M. Protocol for detecting unrecognized sleep apnea in patients with atrial fibrillation by a home-monitoring device: the DAN-APNO study. BMC Cardiovasc Disord. 2022 Jan 8;22(1):6. doi: 10.1186/s12872-021-02453-0. PMID 34998370
- See also: Ectosense - NightOwl device — https://www.ectosense.com